CLINICAL TRIAL: NCT01950325
Title: VRC 601: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC HIVMAB060-00-AB (VRC01), With Broad HIV-1 Neutralizing Activity, Administered Intravenously or Subcutaneously to HIV-Infected Adults
Brief Title: VRC 601: A Phase I, Open-Label, Dose-Escalation Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, VRC HIVMAB060-00-AB (VRC01), With Broad HIV-1 Neutralizing Activity, Administered Intravenously or Subcutaneously to HIV-Infected...
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 130189; 13-I-0189
Record Dates: First submitted 2013-09-21; First posted 2013-09-25 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-08-20

CONDITIONS: HIV-1 Infection; Neutralizing Antibody; Monoclonal Antibody; Viral Load; HIV Antibodies
Keywords: HIV-1 Viral Load; CD4 Count; Antiviral; HIV-1 Infection; Broadly Neutralizing Antibody
MeSH Terms: interventions — VRC01 monoclonal antibody

ARMS (4):
- Group 1 (Experimental): 1mg/kg IV
  Interventions: Biological: VRC-HIVMAB060-00-AB
- Group 2 or Group 3 (Experimental): 5 mg/kg IV (Group 2) or 5 mg/kg SC (Group 3)[only portion of the study that is randomized]
  Interventions: Biological: VRC-HIVMAB060-00-AB
- Group 4 (Experimental): 20 mg/kg IV
  Interventions: Biological: VRC-HIVMAB060-00-AB
- Group 5 (Experimental): 40 mg/kg IV
  Interventions: Biological: VRC-HIVMAB060-00-AB

INTERVENTIONS:
Biological: VRC-HIVMAB060-00-AB — VRC01 Human Monoclonal Antibody

SUMMARY:
This is the first clinical trial of the VRC-HIVMAB060-00-AB (VRC01) monoclonal antibody. VRC01 is a broadly neutralizing antibody directed against HIV. This is a dose-escalation study to examine safety, tolerability, dose and pharmacokinetics of VRC01. The hypothesis is that VRC01 will be safe for administration to HIV-1 infected adults by the intravenous (IV) and subcutaneous (SC) routes and will not elicit hypersensitivity reactions. Samples will be collected to learn if VRC01 is detectable in mucosal secretions and blood of participants and how long VRC01 can be detected in the blood after it is given.

Between 15 and 25 HIV-1 infected adults, ages 18-70 years will be enrolled. There are 4 dose escalation groups for IV administration; the doses are 1 mg/kg, 5 mg/kg, 20 mg/kg and 40 mg/kg. There is 1 group for SC administration at 5 mg/kg. Each group is expected to include at least 3 participants. Each participant will receive two infusions of VRC01 with about 1 month between doses. Infusions are administered in an inpatient unit and an overnight stay at the NIH Clinical Center is required. No more than one subject per day per group will receive a first infusion of the VRC01 product by the IV route and no more than one subject per week will receive a first infusion of the product by the SC route. Study participation lasts for 24 weeks. Participant health and effect on CD4 count and HIV viral load will be monitored. Samples will be collected and stored for research purposes.

...

DETAILED DESCRIPTION:
This is the first clinical trial of the VRC-HIVMAB060-00-AB (VRC01) monoclonal antibody. VRC01 is a broadly neutralizing antibody directed against HIV. This is a dose-escalation study to examine safety, tolerability, dose and pharmacokinetics of VRC01. The hypothesis is that VRC 01 will be safe for administration to HIV-1- infected adults by the intravenous (IV) and subcutaneous (SC) routes and will not elicit hypersensitivity reactions. Samples will be collected to learn if VRC01 is detectable in mucosal secretions and blood of participants and how long VRC01 can be detected in the blood after it is given.

Up to 30 HIV-1 infected adults will be enrolled. Adult 18-60 years old will participate in the dose escalation part of the study. There are 4 dose escalation groups for IV administration; the doses are 1 mg/kg, 5 mg/kg, 20 mg/kg and 40 mg/kg. There is 1 group for SC administration at 5 mg/kg. Each dose escalation group is expected to include at least 3 participants. Each participant during the dose escalation part of the study will receive two infusions of VRC01 with about 1 month between doses, with infusions administered in an inpatient unit and an overnight stay at the NIH Clinical Center required. No more than one subject per day per group will receive a first infusion of the VRC01 product by the IV route and no more than one subject per week will receive a first infusion of the product by the SC route. Study participation lasts for 24 weeks for participants who receive two doses. After the dose escalation is completed, about 10 HIV-infected adults, ages 18-70 years old, with detectable viral load will be enrolled to receive one dose of VRC01 at 40 mg/kg IV with follow-up for 12 weeks. Participant health and effect on CD4 count and HIV viral load will be monitored. Samples will be collected and stored for research purposes.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria:

1. Able and willing to complete the informed consent process.
2. 18-60 years old during the dose escalation; 18-70 years old during subsequent enrollment of viremic subjects.
3. HIV infected and clinically stable,Volunteers during the dose escalation part of the study also must be, without changes in ARV status (whether or not taking an ARV regimen) in the 24 weeks prior to enrollment.
4. Criteria for volunteers enrolling during the dose escalation part of the study:

   Plasma viral load (VL) and CD4 count that meet eligibility criteria on at least two measurements performed within the 24 weeks prior to enrollment. The two measurements used for eligibility must have at least 3 days between tests and at least one set of the tests must be performed at the NIH Clinical Center within the 84 days prior to enrollment.

   If not on ARV treatment, the criteria are:

   -VL less than or equal to 50,000 copies/mL and a CD4 count greater than or equal to 400/mcL.

   If on ARV treatment, the criteria are:

   -VL less than or equal to 50 copies/mL and a CD4 count greater than or equal to 350/mcL.

   Note: A viral blip of <400 copies/mL during the 24 weeks prior to enrollment is permitted if preceded and followed by test results showing VL less than or equal to 50 copies/mL on the same ARV regimen.]

   Criteria for viremic volunteers enrolling after dose escalation is complete:

   At least one detectable plasma viral load greater than or equal to 50 copies/mL and at least one CD4 count greater than or equal to 200 cells/mcL within 84 days prior to enrollment.

   Note: Up to 10 viremic subjects will be enrolled but no more than 4 subjects with a screening VL >100,000 copies/mL will receive VRC01. Other subjects must have a screening VL less than or equal to 100,000 copies/mL
5. In general good health and willing to maintain or establish a relationship with a primary health care provider for medical management of HIV infection while participating in the study.
6. Willing to have blood samples collected, stored indefinitely, and used for various research purposes.
7. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
8. Screening laboratory values within 84 days prior to enrollment must meet the following criteria:

   * absolute neutrophil count greater than or equal to 800/mcL
   * platelets greater than or equal to 100,000/mcL
   * hemoglobin greater than or equal to 10.0 gm/dL
   * creatinine less than or equal to 1.31 mg/dL
   * alanine aminotransferase (ALT) less than or equal to 2.5 times ULN

   Female-Specific Criteria:
9. Agrees not to become pregnant from the time of study enrollment until the last study visit. If a woman is sexually active and has no history of hysterectomy or tubal ligation or menopause, she must agree to use a prescription birth control method or a barrier birth control method.
10. Negative Beta-HCG (human chorionic gonadotropin) pregnancy test (urine or serum) on day of enrollment for any women unless she is post-menopause for 24 consecutive months or has undergone a surgical procedure that precludes pregnancy.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Previous receipt of humanized or human monoclonal antibody whether licensed or investigational.
2. Weight >130 kg or <53 kg.
3. Ongoing AIDS-related opportunistic infection (including oral thrush)
4. Active injection drug use or active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
5. History of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis in the 2 years prior to enrollment.
6. Physical finding on examination considered clinically significant such as murmur (other than functional), hepatosplenomegaly, lymphadenopathy or focal neurological deficit.
7. Hypertension that is not well controlled by medication.
8. Breast-feeding.
9. Receipt of other investigational study agent within 28 days prior to enrollment.
10. Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the volunteer.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2013-08-22; Primary Completion 2015-08-20 (Actual); Study Completion 2015-08-20 (Actual)

PRIMARY OUTCOMES:
Adverse events of all severities | From first product admin thru 56 days after last admin
Solicited systemic adverse events | For 3 days after ea product admin
Serious adverse events and new chronic medical conditions requiring ongoing medical management | From first product admin thru Study Week 24

SECONDARY OUTCOMES:
Pharmacokinetics at each dose level | Thru 4 weeks after first dose and thru 8 wks after second dose
Assess whether anti-drug antibody can be detected in study agent recipients | From first product admin thru Study Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Wu X, Yang ZY, Li Y, Hogerkorp CM, Schief WR, Seaman MS, Zhou T, Schmidt SD, Wu L, Xu L, Longo NS, McKee K, O'Dell S, Louder MK, Wycuff DL, Feng Y, Nason M, Doria-Rose N, Connors M, Kwong PD, Roederer M, Wyatt RT, Nabel GJ, Mascola JR. Rational design of envelope identifies broadly neutralizing human monoclonal antibodies to HIV-1. Science. 2010 Aug 13;329(5993):856-61. doi: 10.1126/science.1187659. Epub 2010 Jul 8. PMID 20616233
- [Background] Wu X, Wang C, O'Dell S, Li Y, Keele BF, Yang Z, Imamichi H, Doria-Rose N, Hoxie JA, Connors M, Shaw GM, Wyatt RT, Mascola JR. Selection pressure on HIV-1 envelope by broadly neutralizing antibodies to the conserved CD4-binding site. J Virol. 2012 May;86(10):5844-56. doi: 10.1128/JVI.07139-11. Epub 2012 Mar 14. PMID 22419808
- [Background] Lynch RM, Tran L, Louder MK, Schmidt SD, Cohen M; CHAVI 001 Clinical Team Members; Dersimonian R, Euler Z, Gray ES, Abdool Karim S, Kirchherr J, Montefiori DC, Sibeko S, Soderberg K, Tomaras G, Yang ZY, Nabel GJ, Schuitemaker H, Morris L, Haynes BF, Mascola JR. The development of CD4 binding site antibodies during HIV-1 infection. J Virol. 2012 Jul;86(14):7588-95. doi: 10.1128/JVI.00734-12. Epub 2012 May 9. PMID 22573869
- [Derived] Lynch RM, Boritz E, Coates EE, DeZure A, Madden P, Costner P, Enama ME, Plummer S, Holman L, Hendel CS, Gordon I, Casazza J, Conan-Cibotti M, Migueles SA, Tressler R, Bailer RT, McDermott A, Narpala S, O'Dell S, Wolf G, Lifson JD, Freemire BA, Gorelick RJ, Pandey JP, Mohan S, Chomont N, Fromentin R, Chun TW, Fauci AS, Schwartz RM, Koup RA, Douek DC, Hu Z, Capparelli E, Graham BS, Mascola JR, Ledgerwood JE; VRC 601 Study Team. Virologic effects of broadly neutralizing antibody VRC01 administration during chronic HIV-1 infection. Sci Transl Med. 2015 Dec 23;7(319):319ra206. doi: 10.1126/scitranslmed.aad5752. PMID 26702094